CLINICAL TRIAL: NCT00680277
Title: Vitamin A Value of Spirulina Carotenoids in Humans
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Nestlé Foundation (Other)
Responsible Party: Guangwen Tang, Tufts University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PV2270
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Intrinsically Labeled Spirulina
Keywords: spirulina; carotenoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Dietary Supplement: spirulina ß-carotene
- 2 (Experimental)
  Interventions: Dietary Supplement: spirulina ß-carotene

INTERVENTIONS:
Dietary Supplement: spirulina ß-carotene — an acute dose of spirulina up to 5 g
  Other Names: spirulina VA study
Dietary Supplement: spirulina ß-carotene — vitamin A value of spirulina ß-carotene
  Other Names: spirulina VA study

SUMMARY:
The goal of this protocol is to determine the vitamin A value (equivalence) of spirulina. The investigation will use intrinsically deuterium labeled spirulina and an isotope vitamin A reference dose, 13C10- retinyl acetate (13C10 RAc), in males (n=20). Up to 45 blood samples (10 ml/sample) will be collected from each subject over a two-month period to evaluate the bioavailability and bioconversion of spirulina ß-carotene to vitamin A.

DETAILED DESCRIPTION:
By utilizing novel stable isotope dilution techniques recently developed in our laboratory, we will trace deuterium labeled ß-carotene in intrinsically labeled spirulina, which is harvested from a hydroponic system. In the mean time, we will track 13C10 labeled vitamin A in humans. In this way we will determine absorption of ß-carotene from spirulina matrix and the conversion of the spirulina ß-Carotene to retinol. This will enable us quantitatively determine the vitamin A equivalence of spirulina.

The specific aims of this study are:

1. To determine labeled ß-C blood response kinetics following an acute dose of intrinsically labeled spirulina;
2. To determine labeled retinol blood response from the intrinsically labeled spirulina;
3. To determine 13C10 retinol blood response from the isotope reference material 13C10 retinyl acetate;
4. To determine s spirulina-vitamin A equivalence.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer

Exclusion Criteria:

* Not has GI track problems
* Any medical condition that will affect the intestinal absorption

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2004-04; Primary Completion 2008-12-31 (Actual); Study Completion 2008-12-31 (Actual)

PRIMARY OUTCOMES:
The enrichment of spirulina ß-carotene and its cleavage product vitamin A were tracked after taken the oral dose of intrinsically labeled spirulina. | 51 days

CONTACTS AND LOCATIONS:
Overall Officials: Guangwen Tang, Ph.D., Principal Investigator — USDA Human Nutrition Research Center on Aging, Tufts University
Locations (1):
- USDA Human Nutrition Research Center on Aging, Tufts Uni., Boston, Massachusetts, United States